CLINICAL TRIAL: NCT03350932
Title: Evaluation of the Effect of Sensory Imagination on Choice of Food Portion Size in School-aged Children
Brief Title: Evaluation of the Effect of Sensory Imagination on Food Portion Size in School-aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: INSEAD (Institut européen d'administration des affaires) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PUNCH 2.4 (2016-A00498-43)
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Sensory Imagination
Keywords: sensory imagination; foods

STUDY DESIGN:
Intervention Model Description: Two groups of children will be constituted: the first group, the control group, will have to perform a sensory imagination task about neutral facts. The second group, the "food sensory imagination" group, will have to perform a sensory imagination task foods.
Who Masked: Participant
Masking Description: Children will not be aware about the type of comparison that will be made with the data; and they will not be aware in which group they will participate in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group of children, will have to perform a sensory imagination task about neutral facts before choosing the portion size of a food.
- Food sensory imagination (Experimental): This group, the "food sensory imagination" group, will have to perform a sensory imagination task foods (being the intervention) before choosing the portion size of a food.
  Interventions: Behavioral: Sensory imagination about foods

INTERVENTIONS:
Behavioral: Sensory imagination about foods — In both groups, children will be presented with pictures of items. In the control group, the pictures will represent landscapes at different seasons. In the experimental group, the pictures will represent a variety of foods. In the experimental group, based on the pictures representing a variety of foods, children will have to perform a food sensory imagination task before choosing the portion size of a food.
  Arms: Food sensory imagination

SUMMARY:
The objective of this intervention is to evaluate the effect of sensory imagination (i.e., imagining the sensory properties of an object) on the choice of food portion size in school-aged children. Previous research showed that it may help children to choose smaller portion size. The investigators would like to assess whether this effect can be reproduced with two types of food (one with a high energy-density and one with a low energy-density), and in older children.

DETAILED DESCRIPTION:
School-aged children (8-11 years old) will be included in their usual schools to participate in an afternoon snack, organised according to regular arrangements, during two days separated by one week. On each day, the participants will receive a choice of three portion sizes of a food (small, medium, large), and will be asked to chose one of these portions and to eat it for snack. On one day, the high energy-density food will be offered; and on the other day, the low energy-density food. This will be counterbalanced across participants. Moreover, two groups of children will be constituted: the first group, the control group, will have to perform a sensory imagination task about neutral facts. The second group, the "food sensory imagination" group, will have to perform a sensory imagination task foods.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Children with food allergies
* Children who dislike experimental foods

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
portion size | The measure for the two foods will be conducted one week apart
  choice of a portion size among three sizes (small, medium, large), for two different foods

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Nicklaus, PhD, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornil Y and Chandon P (2016) Pleasure as a Substitute for Size: How Multisensory Imagery Can Make People Happier with Smaller Food Portions. Journal of Marketing Research: October 2016, Vol. 53, No. 5, pp. 847-864. https://doi.org/10.1509/jmr.14.0299
- [Derived] Lange C, Schwartz C, Hachefa C, Cornil Y, Nicklaus S, Chandon P. Portion size selection in children: Effect of sensory imagery for snacks varying in energy density. Appetite. 2020 Jul 1;150:104656. doi: 10.1016/j.appet.2020.104656. Epub 2020 Mar 9. PMID 32165270